CLINICAL TRIAL: NCT03641690
Title: Evolution of Serum and Bronchoalveolar Inflammatory Parameters in Patients With Severe Adult Respiratory Distress Syndrome (ARDS) Without or With Extracorporeal Mechanical Assistance
Brief Title: Serum and Bronchoalveolar Inflammatory Parameters in Patients With Severe Adult Respiratory Distress Syndrome
Acronym: ARDS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2013-ZOGHEIB
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-08

CONDITIONS: H1N1 Influenza
Keywords: pandemic influenza; mortality; ICU
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 27 case: Twenty-seven patients were admitted to the ICU with severe pneumonia and with a high probability of viral infection or a previously confirmed diagnosis received Empirical antimicrobial therapy
  Interventions: Other: Empirical antimicrobial therapy
- 70 control: 70 healthy subjects (HS) among blood donors attending the Regional Center for Blood Transfusion (Lille, France).

INTERVENTIONS:
Other: Empirical antimicrobial therapy — All patients with pulmonary symptoms received empirical antimicrobial therapy with ceftriaxone and rovamycin or levofloxacin on admission and this was subsequently adapted to any documented bacterial infection if positive.
  Groups: 27 case

SUMMARY:
Mannose-binding lectin (MBL) plays an important role in the innate immune response. In addition to activating the complement, MBL can induce cytokine production and contribute to a deleterious inflammatory response with severe A(H1N1)pdm09 virus infection. The aim was to determine if serum MBL levels correlate with the risk of mortality in intensive care units (ICU) patients with A(H1N1)pdm09 infection.

Prospective observational study was performed in ICU patients with acute respiratory distress syndrome due to influenza A(H1N1)pdm09 virus. Demographic characteristics and severity indices were recorded at ICU admission. MBL was assayed from blood drawn at influenza diagnosis within 24-48 h following the ICU admission. Outcomes were compared according to MBL levels.

DETAILED DESCRIPTION:
Mannose-binding lectin (MBL) plays an important role in the innate immune response. In addition to activating the complement, MBL can induce cytokine production and contribute to a deleterious inflammatory response with severe A(H1N1)pdm09 virus infection. The aim was to determine if serum MBL levels correlate with the risk of mortality in intensive care units (ICU) patients with A(H1N1)pdm09 infection.

Prospective observational study was performed in ICU patients with acute respiratory distress syndrome due to influenza A(H1N1)pdm09 virus. Demographic and clinical data at admission and during the ICU stay were recorded from the medical files of each patient and collected in a database to evaluate variables potentially associated with in-hospital mortality. Data baselines were recorded at admission. Mechanical ventilation, extracorporeal membrane oxygenation (ECMO) requirements, and the use of vasopressor drugs were noted during ICU stay. To determine illness severity, SAPSII and SOFA scoring systems were applied to all patients within 24 h of ICU admission.Demographic characteristics and severity indices were recorded at ICU admission. MBL was assayed from blood drawn at influenza diagnosis within 24-48 h following the ICU admission. Outcomes were compared according to MBL levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed moderate-to-severe ARDS defined by the presence of bilateral alveolar images, a PaO2 / FiO2 ratio <200 mmHg and the absence of an obvious cardiac cause, with or without the need for mechanical respiratory support extracorporeal circulation or decarboxylation.
* Patient benefiting from nitric oxide.
* Patient requiring continuous curarization.

Exclusion Criteria:

* Chronic renal insufficiency dialysis.
* Severe hepatic insufficiency.
* Patient under guardianship or curatorship or deprived of liberty.
* "light" ARDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient according to the present invention, has self optimized by a medical report: sedation, curarization, protective ventilation and adapted PEEP, under and without treatment with BAL and blood samples on the dry tube and EDTA in its care can be included in our study.
  At the time of the diagnosis of ARDS, and during the aetiological assessment, one can highlight a blood sample, samples of tubes for the assays of the inflammation.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Levels of serum MBL are associated with mortality in critically ill patients with severe A(H1N1)pdm09 viral pneumonia. | 7days
  The aim of the present study was to determine whether levels of serum MBL are associated with mortality in critically ill patients with severe A(H1N1)pdm09 viral pneumonia. When a patient met criteria for ARDS, the closest residual blood sample taken on the same day was obtained from the central hospital laboratory in the 24-48 h following the intubation or in the acute phase of the viral infection. MBL serum concentrations were assayed by an Oligomer ELISA kit (BioPorto) according to the manufacturer's instructions. Results are expressed as median [interquartile range (IQR)] or number (percent). Survivors were compared with nonsurvivors using the Mann-Whitney U test for continuous variables and Chi2 test for categorical variables with Yates' correction or Fisher's exact test if necessary. A correlation was searched between MBL and inflammatory parameters using spearman test.

CONTACTS AND LOCATIONS:
Overall Officials: Elie ZOGHEIB, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No